CLINICAL TRIAL: NCT06687681
Title: Efficacy of the Intrathecal Injection of Active Allogeneic Natural Killer Cells in Patients With High-grade Gliomas; A Multi-center Phase II Clinical Trial
Brief Title: Injection of Active Allogeneic Natural Killer Cells in Patients With Gliomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marzieh Ebrahimi (Industry)
Responsible Party: Sponsor-Investigator, Marzieh Ebrahimi, Professor of Medical Immunology, Kian Immune Cell Company
Organization: Kian Immune Cell Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.ACECR.ROYAN.REC.1402.001
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioma Glioblastoma Multiforme; High Grade Glioma (III or IV)
Keywords: natural killer cells; Brain glioma; NK cells; glioblastoma; high grade gliomas
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): patients will recieve 3 cources of 2* 10 8 intrathecal infusion of NK cells every 3 weeks
  Interventions: Biological: NK cell therapy
- Control group (No Intervention): patients will recieve only conventional treatment

INTERVENTIONS:
Biological: NK cell therapy — Active NK cell injection through lumbar puncture in patient with Astrocytoma IDH-mutant, Oligodendroglioma IDHmutant, Glioblastoma IDH-wild type, Diffuse midline glioma, Diffuse hemispheric glioma, Diffuse pediatrictype high-grade glioma IDH-wild type
  Arms: Test group

SUMMARY:
Gliomas are the most common malignant brain tumors, which are often associated with high-grade tumors characterized by an inferior prognosis and low patient survival rates in both children and adults. Surgical removal and tumor resection are the primary treatment approaches for gliomas. In such cases, whole-brain radiation therapy is also employed as a therapeutic option, which itself has significant side effects, and studies have shown limited impact on improving patient survival. Targeted therapy and recently investigated approaches such as targeted therapy have shown some tumor regression, but in most cases, tumor recurrence has been observed after initial regression. Therefore, they have a limited impact on prolonging patient survival. Immunotherapy, particularly immunotherapy with specific immune cells, can effectively identify and eliminate cancer cells and has been utilized as a new approach in the past two decades, especially in cancers where conventional methods have limited success. Among the effective immunotherapy methods, using natural killer cells (NK cells) can be one of the promising approaches. Currently, phase I clinical trials have been conducted by our research group in patients with gliomas.

DETAILED DESCRIPTION:
Inclusion criteria:

New diagnosed patients with grade 3 or 4 brain tumor, based on WHO classification, which are included in the one of the following conditions: • Astrocytoma, IDHmutant • Oligodendroglioma, IDH-mutant • Glioblastoma, IDH-wild type • Diffuse midline glioma • Diffuse hemispheric glioma • Diffuse pediatric-type high-grade glioma, IDH-wild type Age range of 3 to 60 years old both sex Lansky/Karnofsky performance score above 60 Obtained informed consent of patients or parents or legal attendance in cases of pediatrics Hemoglobin above 10 gr/dL of blood Absolute granulocyte count (AGC) above 500 per microliter of blood Platelet count above 50000 per microliter of blood INR below 2 and PTT less than 1.5 times of maximum normal value Plasma bilirubin level less than 1.5 times of maximum normal value Plasma hepatic transaminases (ALT and AST) level less than 3 times of maximum normal value Plasma creatinine level less than 1.5 times of maximum normal value

Exclusion criteria:

Evidence of radio necrosis in MRI or MRS Intolerance of new treatment due to emergency condition History of other malignancies History of any immunodeficiency diseases or any immune compromising conditions Rupture of cerebral shunt or unable to perform a lumbar puncture Pregnancy History of uncontrolled chronic diseases such as: Diabetes, CHF, liver cirrhosis, CKD, etc

ELIGIBILITY:
Inclusion Criteria: New diagnosed patients with grade 3 or 4 brain tumor, based on WHO classification, which are included in the one of the following conditions: • Astrocytoma, IDHmutant • Oligodendroglioma, IDH-mutant • Glioblastoma, IDH-wild type • Diffuse midline glioma • Diffuse hemispheric glioma • Diffuse pediatric-type high-grade glioma, IDH-wild type Age range of 3 to 60 years old both sex Lansky/Karnofsky performance score above 60 Obtained informed consent of patients or parents or legal attendance in cases of pediatrics Hemoglobin above 10 gr/dL of blood Absolute granulocyte count (AGC) above 500 per microliter of blood Platelet count above 50000 per microliter of blood INR below 2 and PTT less than 1.5 times of maximum normal value Plasma bilirubin level less than 1.5 times of maximum normal value Plasma hepatic transaminases (ALT and AST) level less than 3 times of maximum normal value Plasma creatinine level less than 1.5 times of maximum normal value -

Exclusion Criteria: Evidence of radio necrosis in MRI or MRS Intolerance of new treatment due to emergency condition History of other malignancies History of any immunodeficiency diseases or any immune compromising conditions Rupture of cerebral shunt or unable to perform a lumbar puncture Pregnancy History of uncontrolled chronic diseases such as: Diabetes, CHF, liver cirrhosis, CKD, etc

-

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
To measure tumor response after infusion of intrathecal NK cells | From enrollment to the end of treatment at 12 months
  Imaging and Immunotherapy Response Assessment in Neuro-oncology (iRANO) guidelines

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment to the end of treatment at one months
  Using CTCAEs (Common Terminology Criteria for Adverse Events) checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Rasoul Akram hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No